CLINICAL TRIAL: NCT05447247
Title: Clinical Study on Treatment of Neurogenic Bladder by Electroacupuncture on Ba Liao Point Under Ultrasound Guidance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QiluH-xinshenglianhua
Record Dates: First submitted 2022-07-03; First posted 2022-07-07 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-05

CONDITIONS: To Investigate the Clinical Effect of Acupuncturing Ba Liao for Neurogenic Bladder Under the Guidance of Ultrasound

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncturing Ba Liao point under ultrasound guidance (Experimental)
  Interventions: Other: Acupuncturing Ba Liao point under ultrasound guidance
- Conventional acupuncture (Experimental)
  Interventions: Other: Acupuncturing Ba Liao point under ultrasound guidance

INTERVENTIONS:
Other: Acupuncturing Ba Liao point under ultrasound guidance — Acupuncturing Ba Liao point under ultrasound guidance

SUMMARY:
To explore acupuncture under the premise of real-time, dynamic and accurate positioning of Ba liao point with ultrasound, observe the clinical efficacy of treating neurogenic bladder, clarify the essence of acupoints, and provide a new method for the standardization of acupuncture and moxibustion.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis of neurogenic bladder conforms to the main points;
2. Symptoms and signs: patients with lower urinary tract dysfunction such as frequency of urination, urgency of urination, inadequacy of urine or retention of urine, urinary incontinence; Physical examination showed paresthesia in perineum and saddle area.
3. Auxiliary examination; Routine urine examination, B - ultrasonography of urinary system and urodynamic examination.
4. Indwelling catheter has been removed;
5. Conscious and able to accurately express symptoms and signs;
6. Patients who inform patients and their families of the research situation in detail and obtain their consent for treatment.

   -

Exclusion Criteria:

1. Lower urinary tract dysfunction caused by non-nervous system factors such as urethral calculi and organic obstruction;
2. patients with serious heart and lung diseases, liver and hematopoietic diseases and mental diseases;
3. patients with prostate cancer, urethral stricture, bladder neck fibrosis, interstitial cystitis, glandular cystitis and other diseases;
4. patients implanted with urethral stents or sacral nerve electrodes;
5. pregnant and lactation women;
6. Fear of acupuncture, needle-sickness and blood sickness. -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Urodynamic study | Once every two weeks:Before treatment, two weeks after treatment, four weeks after treatment
  Residual urine volume, maximum urine flow rate, average urine flow rate, urination time, urine flow time and urine flow rate were assessed
Neurogenic bladder symptom score | Once every two weeks:Before treatment, two weeks after treatment, four weeks after treatment.followed up for 3 months after treatment
  Patients were evaluated for neurogenic bladder symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China